CLINICAL TRIAL: NCT01089959
Title: The Effect of Esomeprazole 40 mg. Daily for 7 Days on Acid Reflux and Related Arousals During Sleep in Patients With Gastroesophageal Reflux Disease (GERD).
Brief Title: Effect of Esomeprazole 40 mg.Daily for 7 Days on Acid Reflux and Related Arousals During Sleep in Patients With GERD
Acronym: ISS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: RONNIE FASS M.D., SOUTHERN AZ. VA HEALTH CARE SYSTEM
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISS Astra Zeneca 7 day Nexium
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Acid re-flux,GERD; sleep related arousals due to GERD; Treatment of acid reflux during sleep in patients with GERD.
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esomeprazole (Other): Effect of PPI esomeprazole on acid reflux & related arousals during sleep in patients with GERD.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — 40 mg daily for 7 days
  Other Names: Nexium
Drug: esomeprazole — 40 mg. daily, oral medication, once daily for 7 days.
  Other Names: Nexium

SUMMARY:
The purpose of this study is to determine if esomeprazole 40 mg. once daily improves not only nighttime symptoms but also significantly reduces conscious awakenings associated with gastroesophageal reflux and consequently improves sleep quality.

DETAILED DESCRIPTION:
Twenty GERD patients with nighttime heartburn and/or regurgitation at least 3 times a week will be invited to participate in the study. All patients will undergo upper endoscopy to determine presence or absence of esophageal inflammation(using Los Angeles criteria). All patients will be evaluated by the Demographic,Berlin,Epworth Sleepiness Scale Questionnaires, and GERD Symptom Checklist. Thereafter,patients will undergo pH testing w/ an actigraph.The morning of pH probe removal,a Sleep Quality Questionaire will be administered.

Subjects will then receive esomeprazole 40 mg. once daily(30 minutes before breakfast) for 1 week. On day 7,subjects will again undergo pH testing w/ actigraphy, and the results will be analyzed again w/ new integrative software. On the morning of pH probe removal, the sleep Quality Questionnaire will be re-administered.

ELIGIBILITY:
Inclusion Criteria:

* Nocturnal symptoms at least twice a week.
* Ages 18-80
* Erosive esophagitis and/or abnormal pH test -
* Able to read, understand, and complete study questionnaires

Exclusion Criteria:

* Subjects with Barrett's esophagus or peptic stricture on endoscopy
* Subjects with normal endoscopy and pH test
* Subjects with previous upper gastrointestinal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The Effect of Esomeprazole 40 mg. Daily for 7 Days on Acid Reflux and Related Arousals During Sleep in Patients w/ GERD. | 2 years
  This is the first study to evaluate the impact of antireflux treatment, not only on heartburn during sleep, but also on reflux-related conscious awakenings.
  This has not been done previously and will thus provide an opportunity to assess the impact of esomeprazole on nighttime symptoms and awakenings.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — SAVAHCS
Locations (1):
- Southern Arizona VA Health Care System, Tucson, Arizona, United States